CLINICAL TRIAL: NCT05508919
Title: Effect of EMG, RESP, and TEMP Biofeedback Training to Reduce Anxiety Among Undergraduate Students
Brief Title: Effect of Biofeedback Training to Reduce Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Karachi (Other)
Collaborators: Advanced Education & Research Center (Other)
Responsible Party: Principal Investigator, Shamoon Noushad, University of Karachi, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTRA2022
Record Dates: First submitted 2022-06-28; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Anxiety
Keywords: Biofeedback Training; Anxiety; Nursing Students; EMG; Respiration; Temperature
MeSH Terms: conditions — Anxiety Disorders; Respiratory Aspiration | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback Group (Experimental): * The training consists of a total of 8 sessions for every individual with 2 sessions per week over the duration of 4 weeks. Each session will be approximately of 1 to 1.30 hour.
  * Subjects will be given clear instructions to not to use chocolate, coffee, tea and cocoa drinks at least 3 hours before the training session.
  * Since it is suggested that Anxiety tends to change with time so we might consider a one-month pretreatment measure as well as a just before treatment measure. That way we can be sure if our baseline is stable or not.
  * Baseline session: Subject will be asked to sit quietly for 15 minutes and their breathing rate, skin temperature and muscle tension using EMG will be measure without giving any intervention.
  * Subjects will then be given biofeedback training gradually to control their breathing rate, relaxed their muscle activity and temperature through RESP biofeedback, assisted EMG biofeedback and TEMP biofeedback, from the 1st session till their 8th Session.
  Interventions: Device: Biofeedback
- Active Control Group (Active Comparator): Active Control: Writing Sessions The subjects will be asked to take three 20-minute writing sessions and write about the given control topic about their daily events of the past week. For example, in Session 1, we may ask the Subjects to write about how they will use their time. Similarly, we will ask the subject to give more detail and write briefly about the given control condition in session 2 and session 3. At the end of three writing session, we will measure their EMG, RESP and TEMP to compare with the Biofeedback training group.
  Interventions: Other: Writing Sessions

INTERVENTIONS:
Device: Biofeedback — EMG, RESP, and TEMP Biofeedback Training
  Arms: Biofeedback Group
Other: Writing Sessions — The subjects will be asked to take three 20-minute writing sessions and write about the given control topic about their daily events of the past week
  Arms: Active Control Group

SUMMARY:
This study is planned to investigate the effectiveness of EMG, RESP, and TEMP Biofeedback Training to reduce symptoms of anxiety among the nursing students from one school, and to determine whether biofeedback training is associated to relax the minds and bodies of the anxious nursing students to cope with the distressing situation. Study subjects meeting the eligibility criteria will be randomized into two groups using randomly generated numbers: the Biofeedback training group and Control group. Biofeedback training will be used as an intervention vs the control. All the study subjects providing the consent to participate will be made to complete the study questionnaires (Demographic, Screening for Anxiety using the State-Trait Anxiety Inventory -STAI) at baseline and at post-intervention (after 4 weeks).

DETAILED DESCRIPTION:
Study Design:

This study will be conducted as a randomized control trial using subjects from one nursing school. Study subjects meeting the eligibility criteria will be randomized into two groups; the Biofeedback training group receiving EMG, RESP, and TEMP Biofeedback Training, and the Control group in which subjects will be asked to take three 20-minute writing sessions and write about the given control topic about their daily events of the past week. All the study subjects providing the consent to participate will be made to complete the study questionnaires (Demographic, Screening for Anxiety using the State-Trait Anxiety Inventory -STAI6, 7) at baseline and at post-intervention (after 4 weeks).

Study participants will be recruited from the School of Nursing, Koohi Goth Women Hospital, Karachi-Pakistan. Our targeted population will be students from diverse ethnicity and will be considered eligible for participation if they indicated to have anxiety in the pre-screening using the anxiety scale. Students will be invited to take part in the study through advertisement representation on the notice board of the institute. Written informed consent will be obtained from each enrolled subject after providing detail regarding the objectives, duration, and purpose of the study.

Interventions:

The experimental intervention (EMG, RESP, and TEMP Biofeedback):

For this study, we will be using the Alive Pioneer with the GP8 Amp. GP8 Amp can record ECG Heart Rate, EMG for muscle tension, Hand Temperature and Skin conductance. Subjects in this group will get EMG, RESP, and TEMP biofeedback intervention training.

Electromyography Biofeedback (EMG) The surface EMG disposable sticky sensors will be attached to the bicep or flexor muscle. The ground sensor will be attached to subjects' fingertips to read the heart rate. A conductive paste, such as Ten20 Conductive Paste, can be used to improve the connection on hairy areas. The electrodes can be placed one right after another. Attach the white, black, and green lines from the GP8 Amp to the disposable electrodes, in order to see the EMG signals.

Respiration Biofeedback (RESP) In this training the GP8 Amp Reparation belt will be used. The Respiration Belt is placed around the abdomen or chest to measure the subject breathing. As the subject breathe, the belt stretches slightly, and this stretch (near the middle of the belt) is measured. The respiration data is shown as a yellow line in the breath pacer area in the Alive Bottom Graphs. The yellow respiration line shows how the subject breathing affects his/her heart rate and smoothness.

Temperature Biofeedback (TEMP) As suggested that temperature in the hand increases when one get relax. Using GP8 Amp, we can teach the subjects to increase their hand temperature dramatically. The temperature sensor is attached to the GP8 Amp in the mini-USB slot nearest the 4 leads. The other end of temperature sensor will be placed in the subject finger, using one of the skin conductance Velcro finger straps to hold the temperature sensor in place. It will take 30 seconds to 1 minute for temperature to calibrate, until the temperature measured stops increasing, then the training begins.

The sequence of the biofeedback training sessions is given below:

1. The training consists of a total of 8 sessions for every individual with 2 sessions per week over the duration of 4 weeks.
2. Each session will be approximately of 1 to 1.30 hour.
3. Subjects will be given clear instructions to not to use chocolate, coffee, tea and cocoa drinks at least 3 hours before the training session.
4. Since it is suggested that Anxiety tends to change with time so we might consider a one-month pretreatment measure as well as a just before treatment measure. That way we can be sure if our baseline is stable or not.
5. Baseline session: Subject will be asked to sit quietly for 15 minutes and their breathing rate, skin temperature and muscle tension using EMG will be measure without giving any intervention.
6. Subjects will then be given biofeedback training gradually to control their breathing rate, relaxed their muscle activity and temperature through RESP biofeedback, assisted EMG biofeedback and TEMP biofeedback, from the 1st session till their 8th Session.

The control intervention:

In control intervention, the subjects will be asked to take three 20-minute writing sessions and write about the given control topic about their daily events of the past week. For example, in Session 1, we may ask the Subjects to write about how they will use their time. Similarly, we will ask the subject to give more detail and write briefly about the given control condition in session 2 and session 3. At the end of three writing session, we will measure their EMG, RESP and TEMP to compare with the Biofeedback training group.

At the end of biofeedback training and writing sessions, the participants of both groups will also be asked to again fill the State-Trait Anxiety Inventory -STAI scale.

ELIGIBILITY:
Inclusion Criteria:

* Subject must not have any evidence of any metastatic disease.
* Subject must be able to properly write and speak Urdu or English Language.
* Subject must be a first- or second-year student.
* Subject should have high anxiety that will be assessed using the State-Trait Anxiety Inventory-STAI.

Exclusion Criteria:

* Subjects with any history of anxiolytic, antidepressant or other psychiatric medications will be excluded.
* Subjects with any codified psychiatric disorder will be excluded.
* Subjects who smoke or used alcohol will be excluded.
* Subjects who received any structured psychological intervention, psychotherapy or biofeedback or relaxation training will be excluded.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Effective Biofeedback Training | 4 Weeks
  Biofeedback will be demonstrated as a possible effective and useful technique in helping individuals with anxiety over the duration of training of 4 weeks using he State-Trait Anxiety Inventory -STAI at baseline and post-intervention

SECONDARY OUTCOMES:
Electromyography (EMG) | 4 Weeks
  Over the duration of training of 4 weeks, study subjects will be trained to decrease EMG using EMG Biofeedback
Respiratory Rate | 4 Weeks
  Over the duration of training of 4 weeks, study subjects will be trained to decrease Respiratory Rate
Temperature | 4 Weeks
  Over the duration of training of 4 weeks, study subjects will be trained to increase their Skin Temperature

CONTACTS AND LOCATIONS:
Overall Officials: Shamoon Noushad, PhD, Principal Investigator — University of Karachi
Locations (1):
- Koohi Goth Women Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chalo P, Pereira A, Batista P, Sancho L. Brief Biofeedback Intervention on Anxious Freshman University Students. Appl Psychophysiol Biofeedback. 2017 Sep;42(3):163-168. doi: 10.1007/s10484-017-9361-5. PMID 28527121
- [Result] Ratanasiripong P, Ratanasiripong N, Kathalae D. Biofeedback Intervention for Stress and Anxiety among Nursing Students: A Randomized Controlled Trial. ISRN Nurs. 2012;2012:827972. doi: 10.5402/2012/827972. Epub 2012 Jun 28. PMID 22811932
- [Result] Gholami Tahsini Z, Makvand Hosseini S, Kianersi F, Rashn S, Majdara E. Biofeedback-Aided Relaxation Training Helps Emotional Disturbances in Undergraduate Students Before Examination. Appl Psychophysiol Biofeedback. 2017 Dec;42(4):299-307. doi: 10.1007/s10484-017-9375-z. PMID 28761991
- [Result] McAusland L, Addington J. Biofeedback to treat anxiety in young people at clinical high risk for developing psychosis. Early Interv Psychiatry. 2018 Aug;12(4):694-701. doi: 10.1111/eip.12368. Epub 2016 Aug 29. PMID 27573093
- [Result] Niles AN, Haltom KE, Mulvenna CM, Lieberman MD, Stanton AL. Randomized controlled trial of expressive writing for psychological and physical health: the moderating role of emotional expressivity. Anxiety Stress Coping. 2014 Jan;27(1):1-17. doi: 10.1080/10615806.2013.802308. Epub 2013 Jun 6. PMID 23742666
- [Result] Schoenberg PL, David AS. Biofeedback for psychiatric disorders: a systematic review. Appl Psychophysiol Biofeedback. 2014 Jun;39(2):109-35. doi: 10.1007/s10484-014-9246-9. PMID 24806535
- [Result] Prato CA, Yucha CB. Biofeedback-assisted relaxation training to decrease test anxiety in nursing students. Nurs Educ Perspect. 2013 Mar-Apr;34(2):76-81. doi: 10.5480/1536-5026-34.2.76. PMID 23763019